CLINICAL TRIAL: NCT05219682
Title: Changes in Brain Activity in Tactile Stimulus Therapy and Ruka Ruk Therapy Compared to Mirror Therapy in Upper Limb Rehabilitation.
Brief Title: Changes in Brain Activity During Mirror Therapy and Virtual Reality Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Kateřina Pilátová, Bc., Charles University, Czech Republic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 200/2020
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Healthy; Age of Probands 18 - 55 Years
Keywords: EEG; Virtual Reality; Rehabilitation; Mirror neurons; Mirror Therapy
MeSH Terms: interventions — Mirror Movement Therapy; Rehabilitation

STUDY DESIGN:
Intervention Model Description: Each participant started with EEG measurements at rest followed by 3 EEG measurements in mirror therapy and 3 EEG measurements with mirror therapy in virtual reality. The order of measurement was randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: electroencephalographic measurement — recording brain activity in mirror therapy, haptic and tactile stimulation and in mirror therapy using virtual reality
  Other Names: Haptic stimulation; tactile foam roller stimulation; mirror therapy; Virtual reality; Rehabilitation

SUMMARY:
The purpose of this study is to compare electroencephalographic activity in upper limb rehabilitation with mirror therapy and virtual reality rehabilitation.

DETAILED DESCRIPTION:
This is an experiment measuring EEG to healthy adult probands during mirror therapy and VR mirroring therapy in the upper limb. The experiment will be supplemented by haptic contact and stimulation of the upper limb with a foam roller. According to the instructions, the participants will perform a predetermined movement with one upper limb - clenching the fist. In one part with the mirror, in the other part the sensor for sensing the movement of the hand detects the movement, the software creates the illusion that the patient performs the same movement with the dominant and non-dominant upper limb. The patient sees on the screen the illusion of movement of both of his upper limbs. During therapy, the other upper limb will be tactively stimulated haptically and with a foam roller. Data collection will take place by measuring the electrical activity of the brain using an EEG device. The obtained data will then be processed and evaluated with the help of the sLORETA program. The aim of this work is to compare the brain activity from the above therapies with the resting state of the proband and to focus on the activity of mirror neurons.

ELIGIBILITY:
Inclusion Criteria:

* a healthy individual with a valid medical examination.

Exclusion Criteria:

* Having a stroke or other illness that is related to a disorder of movement of the upper limbs. Severe visual or auditory deficit and decompensated epilepsy due to screen movement tracking. Persons with acute (especially infectious) diseases did not participate in the research.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of EEG for each intervention versus the resting phase of the measurement | month
  After processing the data in the sLORETA program, statistically significant places with different brain activity during interventions were identified, each type of intervention is evaluated separately.

SECONDARY OUTCOMES:
Comparison of electroencephalographic recordings from mirror therapy with therapy in virtual reality | month
  After processing the data in the sLORETA program, statistically significant places with different brain activity during interventions were identified, each type of intervention is evaluated separately.

CONTACTS AND LOCATIONS:
Overall Officials: MUDr. David Pánek, Ph.D., Study Director — Employee
Locations (1):
- Faculty of Physical Education and Sport at Charles University, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided